CLINICAL TRIAL: NCT00706745
Title: Possible Effects of Supplementation With Cis-9, Trans-11 Conjugated Linoleic Acid on Markers of Atherosclerosis
Brief Title: Conjugated Linoleic Acid and Atherosclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: University of Aberdeen (Other); Lipid Nutrition B.V (Unknown); Center Novem (Unknown)
Responsible Party: Principal Investigator, Michiel L. Bots, Professor of Epidemiology of Cardiovascular Disease, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLA362
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; dietary supplements; randomised controlled trial; arterial stiffness; linoleic acid
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): The control oil is based on the general fat consumption in a Western population and consists of an equal amount (4 gr) of fat. It is a blend of palm (80%) and soybean oil (20%). Two capsules will be taken in the morning and two in the evening.
  Interventions: Dietary Supplement: oil rich in cis9, trans11 conjugated linoleic acid; Dietary Supplement: placebo
- oil rich in cis9, trans11 CLA (Active Comparator): Subjects will receive daily 4 g of CLA oil (2.6 g cis9,trans11-CLA), 2 capsules to be taken in the morning and 2 in the evening.
  Interventions: Dietary Supplement: oil rich in cis9, trans11 conjugated linoleic acid; Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: oil rich in cis9, trans11 conjugated linoleic acid — An oil rich in cis9, trans11 conjugated linoleic acid (cis9,trans11-CLA). Of the total amount of CLA in the oil, 80% is cis9, trans11-CLA and 20% trans10, cis12-CLA. In total 4 grams of oil will be given daily. The oil will be taken in the form of soft gel capsules. Two capsules will be taken in the morning and two in the evening.
  Other Names: oil rich in cis9, trans11 CLA
Dietary Supplement: placebo — identical placebo capsules.
  Other Names: no other names

SUMMARY:
Rationale: Cis-9, trans-11 conjugated linoleic acid (CLA) can protect against the atherosclerosis development in several animal models. Studies in transgenic mice have shown that mechanisms might involve beneficial effects on lipoprotein metabolism and insulin sensitivity and in addition activation of anti-inflammatory pathways. A very limited amount of human studies have not shown similar beneficial effect of cis9,trans11-CLA on insulin sensitivity in obese subjects, yet cis9,trans11-CLA did improve the lipoprotein profile in healthy subjects. The effect of cis9,trans11-CLA supplementation on alternative early biomarkers of atherosclerosis, like aortic pulse wave velocity, and alternative biomarkers identified through platelet proteomics, has not been assessed before, and may add valuable insights into the mechanism of this functional fatty acid in humans.

Objective: To assess the effect of increased intake of cis9 trans11-CLA on development of atherosclerosis, as assessed with aortic pulse wave velocity and on alternative biomarkers.

Study design: The study is designed as a double blind randomised placebo controlled parallel group trial.

Study population: 400 men and women, between 40 and 70 years of age, with a body mass index of 25 kg/m2 or above. Subjects with previous symptomatic vascular disease or diabetes mellitus and subjects on blood pressure lowering or lipid lowering medication are excluded.

Intervention: Subjects in the intervention arm will receive daily 4 g of CLA oil (2.6 g cis9,trans11-CLA), 2 capsules to be taken in the morning and 2 in the evening. The subjects in the control arm receive 4 identical placebo capsules.

Main study parameters/endpoints: The main study outcome is difference between treatment arms in change in aortic pulse wave velocity after 6 months intervention.

DETAILED DESCRIPTION:
Rationale: Cis-9, trans-11 conjugated linoleic acid (CLA) can protect against the atherosclerosis development in several animal models. Studies in transgenic mice have shown that mechanisms might involve beneficial effects on lipoprotein metabolism and insulin sensitivity and in addition activation of anti-inflammatory pathways. A very limited amount of human studies have not shown similar beneficial effect of cis9,trans11-CLA on insulin sensitivity in obese subjects, yet cis9,trans11-CLA did improve the lipoprotein profile in healthy subjects. The effect of cis9,trans11-CLA supplementation on alternative early biomarkers of atherosclerosis, like aortic pulse wave velocity, and alternative biomarkers identified through platelet proteomics, has not been assessed before, and may add valuable insights into the mechanism of this functional fatty acid in humans.

Objective: To assess the effect of increased intake of cis9 trans11-CLA on development of atherosclerosis, as assessed with aortic pulse wave velocity and on alternative biomarkers.

Study design: The study is designed as a double blind randomised placebo controlled parallel group trial.

Study population: The study population comprises 400 men and women, between 40 and 70 years of age, with a body mass index of 25 kg/m2 or above. Subjects with previous symptomatic vascular disease or diabetes mellitus and subjects on blood pressure lowering or lipid lowering medication are excluded.

Intervention: Subjects in the intervention arm will receive daily 4 g of CLA oil (2.6 g cis9,trans11-CLA), 2 capsules to be taken in the morning and 2 in the evening. The subjects in the control arm receive 4 identical placebo capsules.

Main study parameters/endpoints: The main study outcome is difference between treatment arms in change in aortic pulse wave velocity after 6 months intervention. Secondary outcomes are differences between treatment groups in change in serum lipids (total, LDL- and HDL cholesterol and triglycerides) and change in systolic and diastolic blood pressure, as well as in F2-isoprostanes and platelet biomarkers of haemostatic function (proteomics). Blood samples will be stored for assessment of plasma parameters of glucose intolerance, inflammation and endothelial function.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The assessment of aortic pulse wave velocity is non-invasive and does not carry any risks nor has any side effects. The assessment of lipids and blood pressure might sometimes carry some discomfort but can be seen as routine procedures. Completion of questionnaire needs to done once. The participants need to come to the research center three times. Based on findings of several short-term and long-term studies using the compound, no excess serious adverse events were found.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent
* Healthy men and women
* Between 40-70 years of age
* Body mass index > 25 kg/m2

Exclusion Criteria:

* Inability to understand the patient information
* Inability to speak, read and understand the Dutch language
* Indication (BP over 160/90) or using blood pressure lowering drugs
* Indication (total cholesterol > 8 mmol/l) or using lipid lowering drugs
* Indication (glucose > 7 mmol/l) or using glucose lowering drugs
* Alcohol abuse (>21 alcoholic beverages per week)
* Women who are pregnant, lactating or who are planning to become pregnant
* Symptomatic vascular disease
* Use of fish oils (omega 3/6,capsules or oil)
* Use of plant stanols/sterols (margarines like benecol, pro active)
* Use of weight loss supplements
* Receipt of any investigational treatment (drug or device) within 30 days prior to visit 1

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The main study outcome is difference between treatment arms in change in aortic pulse wave velocity after 6 months intervention. | 6 months

SECONDARY OUTCOMES:
change in serum lipids (total, LDL- and HDL cholesterol and triglycerides) and change in systolic and diastolic blood pressure and platelet biomarkers of haemostatic function (proteomics). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michiel L Bots, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- Julius Center for Health Sciences and Primary Care, UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] Sluijs I, Plantinga Y, de Roos B, Mennen LI, Bots ML. Dietary supplementation with cis-9,trans-11 conjugated linoleic acid and aortic stiffness in overweight and obese adults. Am J Clin Nutr. 2010 Jan;91(1):175-83. doi: 10.3945/ajcn.2009.28192. Epub 2009 Nov 18. PMID 19923377
- [Result] Bachmair EM, Bots ML, Mennen LI, Kelder T, Evelo CT, Horgan GW, Ford I, de Roos B. Effect of supplementation with an 80:20 cis9,trans11 conjugated linoleic acid blend on the human platelet proteome. Mol Nutr Food Res. 2012 Jul;56(7):1148-59. doi: 10.1002/mnfr.201100763. Epub 2012 May 30. PMID 22648731